CLINICAL TRIAL: NCT00933673
Title: Phase II Study of L-asparaginase Plus DICE Regimen in Patients With Stage I/II NK/T-cell Lymphoma
Brief Title: New Combination Regimen of L-asparaginase, Dexamethasone, Ifosfamide, Cisplatin and Etoposide in NK/T-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 09-02
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Lymphoma
Keywords: NK/T cell lymphoma; DICE; L-asparaginase
MeSH Terms: conditions — Lymphoma; Lymphoma, Extranodal NK-T-Cell | interventions — Asparaginase; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-DICE (Experimental)
  Interventions: Drug: L-asp, DXM, IFO, VP-16, DDP

INTERVENTIONS:
Drug: L-asp, DXM, IFO, VP-16, DDP — L-asp 6000 u/m2; DXM 40 mg d1-4; IFO 1200mg/m2 d1-4; Mesna 400mg, tid, d1-4; VP-16 60 mg/m2 d1-4; DDP 20mg/m2 d1-4; q3w. Efficacy was evaluated every two cycles. If patients hadn't diseases progression, two more cycles and radiation would be administered.
  Other Names: L-DICE

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the combination chemotherapy of L-asparaginase plus DICE regimen in the patients with early stage NK/T-cell lymphoma.

DETAILED DESCRIPTION:
DICE regimen was found to be highly effective as induction chemotherapy in patients with early stage NK/T-cell lymphoma in the ongoing study. L-asparaginase, an agent with unique anti-cancer mechanism, was also found to be effective in salvage setting. In terms of non-overlapped efficacy and toxicity, the investigators designed this phase II study to verify the efficacy and tolerability of this new combination.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-75 years old
* Histological confirmed, previously untreated stage I/II NK/T cell lymphoma in the upper-aerodigestive tract
* ECOG performance status less than 2
* Life expectancy of more than 3 months
* Normal laboratory values: hemoglobin > 80 g/dl, neutrophil > 2×109/L, platelet > 100×109/L, serum creatine < 1.5×upper limitation of normal (ULN), serum bilirubin < 1.5×ULN, ALT and AST < 2.5×ULN

Exclusion Criteria:

* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* The evidence of CNS metastasis
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 6 weeks

SECONDARY OUTCOMES:
Overall response rate, PFS and OS | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China